CLINICAL TRIAL: NCT01085812
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Relapse-Prevention Study With F2695 SR in Patients With Major Depressive Disorder
Brief Title: Relapse-Prevention Study With Levomilnacipran ER (F2695 SR) in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVM-MD-05
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): 40, 80 or 120 mg/day Levomilnacipran ER capsules, oral administration, once daily dosing.
  Interventions: Drug: Levomilnacipran ER
- 1 (Placebo Comparator): Matching placebo capsules, oral administration, once daily dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levomilnacipran ER — Drug: Levomilnacipran ER (40, 80 or 120 mg/day) Study drug is to be given orally, in capsule form, once daily.
  Arms: 2
Drug: Placebo — Matching placebo to be given orally, in capsule form, once daily.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Levomilnacipran ER relative to placebo in the prevention of depression relapse in patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
Patients who demonstrate improvement in depressive symptoms at the end of the initial 12-week open-label treatment period with Levomilnacipran ER are randomized to continue Levomilnacipran ER or switch to placebo under double-blind conditions for up to 24 weeks of additional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-65 years old
* Currently meet the DSM-IV-TR criteria for Major Depressive Disorder
* The patient's current depressive episode must be at least 4 weeks in duration

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not practicing a reliable method of birth control
* Patients with a history of meeting DSM-IV-TR criteria for:

  * any manic or hypomanic episode
  * schizophrenia or any other psychotic disorder
  * obsessive-compulsive disorder
* Patients who are considered a suicide risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Forero, MA, Study Director — Forest Laboratories
Locations (35):
- United States (30):
  - Forest Investigative Site #023, Beverly Hills, California
  - Forest Investigative Site #017, Encino, California
  - Forest Investigative Site #021, Garden Grove, California
  - Forest Investigative Site #025, Newport Beach, California
  - Forest Investigative Site #030, Orange, California
  - Forest Investigative Site #002, San Diego, California
  - Forest Investigative Site #003, Sherman Oaks, California
  - Forest Research Institute #001, Bonita Springs, Florida
  - Forest Investigative Site #015, Fort Myers, Florida
  - Forest Investigative Site #029, Maitland, Florida
  - Forest Investigative Site #005, North Miami, Florida
  - Forest Investigative Site #016, Orlando, Florida
  - Forest Investigative Site #004, South Miami, Florida
  - Forest Investigative Site #014, Atlanta, Georgia
  - Forest Investigative Site #022, Chicago, Illinois
  - Forest Investigative Site #006, Chicago, Illinois
  - Forest Investigative Site #009, Prairie Village, Kansas
  - Forest Investigative Site #013, Baltimore, Maryland
  - Forest Investigative Site #010, Boston, Massachusetts
  - Forest Investigative Site #012, St Louis, Missouri
  - Forest Investigative Site #011, Staten Island, New York
  - Forest Investigative Site #026, Portland, Oregon
  - Forest Investigative Site #008, Bridgeville, Pennsylvania
  - Forest Investigative Site #028, Norristown, Pennsylvania
  - Forest Investigative Site #020, Philadelphia, Pennsylvania
  - Forest Investigative Site #024, Memphis, Tennessee
  - Forest Investigative Site #007, Dallas, Texas
  - Forest Investigative Site #019, San Antonio, Texas
  - Forest Investigative Site #018, Bellevue, Washington
  - Forest Investigative Site #027, Seattle, Washington
- Canada (5):
  - Forest Investigative Site #050, Kelowna, British Columbia
  - Forest Investigative Site #051, Vancouver, British Columbia
  - Forest Investigative Site #052, Sydney, Nova Scotia
  - Forest Investigative Site #055, Chatham, Ontario
  - Forest Investigative Site #053, Ottawa, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited over a 10-month period from March of 2010 to January of 2011 at 36 studies sites, 30 in the United States and 6 in Canada.
Pre-assignment Details: Patients began with a 12-week open-label treatment period, followed by a 24-week double-blind treatment period.
Groups:
- Placebo: Matching placebo capsules, oral administration, once daily dosing.
- Levomilnacipran ER: 40, 80 or 120 mg/day Levomilnacipran ER capsules, oral administration, once daily dosing.
Period: Open-Label Period
Arm/Group | Placebo | Levomilnacipran ER
Started | 0 | 734
Completed | 0 | 494
Not Completed | 0 | 240
Not completed — Adverse Event | 0 | 80
Not completed — Lack of Efficacy | 0 | 26
Not completed — Protocol Violation | 0 | 39
Not completed — Withdrawal by Subject | 0 | 53
Not completed — Lost to Follow-up | 0 | 42
Period: Double-Blind Period
Arm/Group | Placebo | Levomilnacipran ER
Started | 113 | 235
Completed | 92 | 177
Not Completed | 21 | 58
Not completed — Adverse Event | 3 | 8
Not completed — Protocol Violation | 2 | 7
Not completed — Withdrawal by Subject | 11 | 24
Not completed — Lost to Follow-up | 5 | 17
Not completed — Other Reasons | 0 | 2
Period: Double-blind Intent-to-treat Population
Arm/Group | Placebo | Levomilnacipran ER
Started | 112 | 230
Completed | 92 | 174
Not Completed | 20 | 56
Not completed — Adverse Event | 3 | 8
Not completed — Protocol Violation | 2 | 7
Not completed — Withdrawal by Subject | 11 | 22
Not completed — Lost to Follow-up | 4 | 17
Not completed — Positive serum pregnancy test result | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Baseline Participant population is based on the 734 enrolled patients who received at least one dose of open-label treatment.
Groups:
- Open Label Levomilnacipran ER: 40, 80 or 120 mg Levomilnacipran ER capsules, oral administration, once daily dosing.
Arm/Group | Open Label Levomilnacipran ER
Number analyzed (Participants) | 734
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.3)
Age, Customized [Count of Participants; unit: Participants]
  18 years to 19 years | 8
  20 years to 29 years | 151
  30 years to 39 years | 127
  40 years to 49 years | 208
  50 years to 59 years | 186
  60 years to 65 years | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 425
  Male | 309
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 683
  Canada | 51
Weight [Mean (Standard Deviation); unit: kg] | 83.41 (18.43)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms Per Meter Squared] | 28.88 (5.42)

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse (Days)
Description: Number of days until patients meet relapse criteria. Relapse was defined as 1 or more of the following: 1. MADRS total score of at least 22 at 2 consecutive visits 2. Increase of 2 or more points in CGI-I score compared with the CGI-I score at Visit 9 at 2 consecutive visits 3. Premature discontinuation due to insufficient therapeutic response 4. MADRS item 10 score of at least 4
Time Frame: 24 Weeks
Population: The double blind Intent-to-treat population consists of 342 randomized participants who received study drug and were evaluated for the Primary Outcome Measure
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Levomilnacipran ER: 40, 80 or 120 mg Levomilnacipran ER capsules, oral administration, once daily dosing.
Arm/Group | Placebo | Levomilnacipran ER
Number analyzed (Participants) | 112 | 230
Days | NA (NA) — Relapse did not occur within the 24-week time frame of the study | NA (NA) — Relapse did not occur within the 24-week time frame of the study

ADVERSE EVENTS:
Time Frame: Adverse event data was collection over a 20-month period from March 2010 to November 2011 at 36 study sites in the U.S and Canada.
Description: The Serious Adverse Event data presented here is for the safety population. The Other Adverse Event data presented here is for the safety population during the 24 week double-blind treatment period.
Groups:
- Placebo - Double Blind Treatment: Matching placebo capsules, oral administration, once daily dosing.
- Levomilnacipran ER - Double Blind Treatment: 40, 80 or 120 mg Levomilnacipran ER capsules, oral administration, once daily dosing.
Arm/Group | Open Label Levomilnacipran ER | Placebo - Double Blind Treatment | Levomilnacipran ER - Double Blind Treatment
All-Cause Mortality (participants affected / at risk) | 0/734 | 0/112 | 0/233
Serious Adverse Events (participants affected / at risk) | 7/734 | 4/112 | 2/233
Other Adverse Events (participants affected / at risk) | 448/734 | 31/112 | 68/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Levomilnacipran ER (N=734) | Placebo - Double Blind Treatment (N=112) | Levomilnacipran ER - Double Blind Treatment (N=233)
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Troponin I increased (Investigations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Open Label Levomilnacipran ER (N=734) | Placebo - Double Blind Treatment (N=112) | Levomilnacipran ER - Double Blind Treatment (N=233)
Nausea (Gastrointestinal disorders) | 160 | 5 | 13
Headache (Nervous system disorders) | 141 | 11 | 31
Constipation (Gastrointestinal disorders) | 82 | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 80 | 1 | 4
Dizziness (Nervous system disorders) | 78 | 5 | 4
Dry mouth (Gastrointestinal disorders) | 78 | 1 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 27/309 | 1/51 | 1/94
Insomnia (Psychiatric disorders) | 63 | 5 | 5
Heart rate increased (Investigations) | 54 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 51 | 10 | 17
Nasopharyngitis (Infections and infestations) | 25 | 9 | 20

LIMITATIONS AND CAVEATS:
This was a failed study. The lower than expected rate of relapse in the placebo group compromised the projected power to demonstrate a difference between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.